CLINICAL TRIAL: NCT01698411
Title: Study of the Influence of Sleep on Hemodynamic Parameters in Patients With Sleep Disorders
Acronym: HATS
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-57; 2012-A00825-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-07-12; First posted 2012-10-03 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Hypertension; Sleep; Insomnia
Keywords: hypertension; sleep; insomnia
MeSH Terms: conditions — Hypertension; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Several epidemiological studies in large cohorts suggest a strong association between sleep duration, complaint of insomnia and risk of hypertension.These findings suggest an important role of sleep quality in development of hypertension. Principal limitations of these studies are the cross-sectional study design, self-report sleep duration and poor measurement of blood pressure. The investigators propose to study an insomniac population with complete evaluation of quality and quantity of sleep, associated to complete hemodynamic measurement of hypertension.

DETAILED DESCRIPTION:
Hypertension and sleep disorders is a cross sectional study realised in an adult cohort with chronic complain of insomnia. In our study, sleep duration is evaluated by complete evaluation of quality and quantity of sleep: one night PSG, associated with sleep agenda during 3 weeks, actigraphy, and several sleep questionnaires. We join to this sleep evaluation, a complete hemodynamic evaluation with: path way velocity and central BP obtained by tonometry, ambulatory BP measurement (ABBM), and self- BP measurement.

The primary objective of this epidemiological study is to show an increase risk of hypertension when sleep duration is less than 7 hours, with objective measurement of sleep duration and hypertension.

Secondary objectives are to evaluate role of complain of insomnia in the risk of hypertension, and to determine cardiovascular risk in insomnia with hemodynamic explorations.

ELIGIBILITY:
Inclusion Criteria:

* adult with insomnia (6 months or more)

Exclusion Criteria:

* sleep disorders with obstructive apnea

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult with chronic complain of insomnia
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
hypertension | one year
  hypertension is defined by blood pressure obtained with 24 hours ambulatory blood pressure measurement when mean blood pressure is over 135/80 in the day, and 125/70 in the night, or when patient take antihypertensive drugs

SECONDARY OUTCOMES:
hemodynamic measures | one year
  central blood pressure, pathway velocity, blood pressure amplification, visit-to-visit variability of blood pressure, cardiac rhythm variability.

CONTACTS AND LOCATIONS:
Overall Officials: jacques blacher, professor, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- centre du sommeil et de la vigilance, Hotel Dieu, Paris, France